CLINICAL TRIAL: NCT00555451
Title: A Phase I, Double-Blind, Placebo-Controlled, Dose Ranging Study of the Safety, Tolerance, Pharmacokinetics and Potential Activity of HE3286 When Administered Orally to Obese Adult Subjects for 28 Days
Brief Title: Safety, Pharmacokinetics and Potential Activity of HE3286 in Obese Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Harbor Therapeutics (Industry)
Responsible Party: Nanette Onizuka-Handa, Sr. Vice President, Regulatory Affairs and Quality, Hollis-Eden Pharmaceuticals
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HE3286-0102
Record Dates: First submitted 2007-11-06; First posted 2007-11-08 (Estimated); Last update posted 2010-05-13 (Estimated); Status verified 2010-05

CONDITIONS: Insulin Resistance
Keywords: phase I; safety; tolerance; insulin resistance; obese; pharmacokinetics
MeSH Terms: conditions — Insulin Resistance; Obesity | interventions — 17-ethynyl-5-androstene-3, 7, 17-triol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: HE3286 — Dose escalating cohort driven study. 6 planned cohorts.
  1. HE3286 5 mg or placebo QD for 28 days;
  2. HE3286 10 mg (5 mg BID) or placebo BID for 28 days
  3. HE3286 20 mg (10 mg BID) or placebo BID for 28 days
  4. HE3286 40 mg (20 mg BID) or placebo BID for 28 days
  5. HE3286 4 mg (2 mg BID), 20 mg (10 mg BID) or placebo BID for 28 days
  6. HE3286 10mg (5 mg BID) for 28 days (open-label cohort in patients with T2DM)

SUMMARY:
The objectives of this study are to evaluate the safety, tolerance and pharmacokinetics of HE3286 when administered daily for 28 days to obese adult subjects and to assess potential activity of HE3286 to decrease insulin resistance. An open-label cohort of 6 patients with type II diabetes mellitus will be treated at 10 mg (5 mg BID).

DETAILED DESCRIPTION:
HE3286 has a potentially new mechanism of action that may improve the current therapeutic options available to patients with metabolic disorders, inflammatory and autoimmune diseases. In preclinical experiments, HE3286 has shown to have anti-inflammatory activity associated with corticosteroids but without the side effects known with corticosteroid use, such as immune suppression and bone loss. HE3286 has demonstrated glucose-lowering and insulin-enhancing effects in several preclinical mouse and rat models of insulin resistance. In these experiments, HE3286 lowered blood glucose levels and prevented progression of hyperglycemia and HE3286 appeared to enhance insulin sensitivity.

ELIGIBILITY:
Main Inclusion Criteria:

* Males or females between 18 and 65 years of age
* Body mass index for females between 29 and 35 kg/m2 and no more than 37 kgm2 for males
* Fasting blood glucose level < 126 mg/dL at screening
* 2 hour postprandial (following 75 grams glucose) blood glucose between 140 to 200 mg/dL
* Normal thyroid stimulating hormone with or without thyroid replacement therapy
* Fasting triglycerides < 350 mg/dL
* For females of reproductive potential, agree to avoid pregnancy during the study and for 3 months following study completion, have a negative serum and/or urine pregnancy test, and use an acceptable method of birth control
* Non-smoker or has not smoked for 6 months prior to the screening visit
* No history of alcohol abuse within 2 years
* Negative drug screen at screening and baseline
* Stable weight (+/- 5%); no history of weight loss or gain (> 10% body weight)
* Must provide voluntary, written, informed consent prior to screening evaluations
* Must be able to swallow capsules

Main Exclusion Criteria:

* Marked prolongation of QT/QTc interval or history of additional risk factors for Torsades de Pointes at screening or baseline
* Positive for HIV, HAV, HBV or HCV
* History of clinically significant cardiovascular, hepatic, respiratory or renal or endocrine disorders
* History of breast and/or prostate cancer
* Clinically significant neurological or psychiatric condition, uncontrolled hypertension, clinically significant unstable medical abnormality, chronic disease or active, serious clinical infection or condition
* Personal or family member with breast and/or prostate cancer
* Malignancy within past 5 years except for successfully treated basal cell carcinoma of the skin
* Personal and/or family history of venous thromboembolism
* History of stroke and/or heart attack
* Medication prohibited from study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
safety and pharmacokinetics | Duration of the study

SECONDARY OUTCOMES:
To assess the potential activity of HE3286 to decrease insulin resistance | duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Dwight R. Stickney, MD, Study Director — Harbor Therapeutics
Locations (2):
- United States (2):
  - Baton Rouge, Louisiana
  - dgd Research, Inc., San Antonio, Texas